CLINICAL TRIAL: NCT02987582
Title: A Feasibility Study of an Emotion-Focused Mindfulness Group to Enhance Coping and Resilience in Family Medicine Patients Living With Common Mental Illness
Brief Title: A Feasibility Study of an Emotion-Focused Mindfulness Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto Practice Based Research Network (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFM 1
Record Dates: First submitted 2016-10-25; First posted 2016-12-09 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Depression; Anxiety
Keywords: mental health; mindfulness; shame
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emotion-focused mindfulness group (Experimental): 8-week mindfulness group
  Interventions: Behavioral: Emotion-focused mindfulness group

INTERVENTIONS:
Behavioral: Emotion-focused mindfulness group — Intervention The group will run for 8-weeks. Each group session is 2 and a half hours. Half way through the intervention there will be a 5 hour retreat on the weekend. A typical group format includes 20-40 minutes of meditation, followed by 10 minutes of independent journaling. Then group members will have time to report on recollections from meditation and facilitators will provide feedback. There is a break and the second part of the group focuses on a didactic teaching topic. Topics change each week; groups will run between October 2016 and June 2018.

SUMMARY:
Living with symptoms of mental illness is associated with psychosocial impairment as it can affect someone's ability to work, their relationships and level of functioning. This also has high economic costs on a societal level. It has been shown that an increase in self-compassion may result in a secondary benefit of reducing psychological distress, which could offer substantial benefits. There is little empirical data on Emotion Focused Mindfulness (EFM) interventions for the population we are studying. This study aims to address this gap in the literature and practice, thus advancing the field.

DETAILED DESCRIPTION:
Study Design

The proposed study is a non-controlled, open-label, repeated measures intervention study. It is a two year feasibility study.

Procedure:

Recruitment

Participants will be recruited through the Mount Sinai Academic Family Health Team. Patients who experience symptoms of depression and/or anxiety, may be referred by any member of the family health team, self-referrals through the family health team will also be accepted. Patients will be screened for eligibility for the EFM Group by the group facilitators. Patients may participate in the EFM group and refuse to participate in the research study.

When patients agree to participate in the group intervention, patients will then be asked about interest in participating in this research. Group facilitators will provide details about the study. Interested patients are given the consent form to review. The group facilitator leaves the room and the research associate will then come into the room to obtain written consent.

Intervention

The group will run for 8-weeks. Each group session is 2 and a half hours. Half way through the intervention there will be a 5 hour retreat on the weekend. A typical group format includes 20-40 minutes of meditation, followed by 10 minutes of independent journaling. Then group members will have time to report on recollections from meditation and facilitators will provide feedback. There is a break and the second part of the group focuses on a didactic teaching topic. Topics change each week. EFM groups will run between September 2016 and June 2018.

ELIGIBILITY:
Inclusion Criteria:

Must be patient of Mount Sinai Academic Family Health Team

* Adults over the age of 18 years
* Symptoms of depression and anxiety as identified by the patient and/or family physician
* Sufficient English language skills to participate in the group (based on assessment of group facilitators)
* Committed and willing to engage in the group work, such as listening to others, speaking in front of others (based on assessment of group facilitators)

Exclusion Criteria: (each based on assessment by group facilitators)

* Active suicidality
* Severe depression
* Possible alcohol abuse
* High tendency to dissociate
* Personality style that may disrupt group formation processes, participation in interpersonal group processes, and/or developing a meditation practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Scale (SCS) to assess change between baseline, midpoint, group completion and 2 months post group. | Weeks 1, 4, 8 and 2 months post group completion
  26 question self-administered questionnaire

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) to assess change between baseline, midpoint, group completion and 2 months post group. | Weeks 1, 4, 8 and 2 months post group completion
  20 item self-report measure of positive and negative affect
Patient Health Questionnaire - Somatic Anxiety Depression Scale (PHQ-SADS) to assess change between baseline, midpoint, group completion and 2 months post group. | Weeks 1, 4, 8 and 2 months post group completion
  Self-report scales that include the 9 questions for assessing depression; 7 questions for assessing general anxiety; and 15 questions for assessing somatic symptoms
Internalized Shame Scale to assess change between baseline, midpoint, group completion and 2 months post group. | Weeks 1, 4, 8 and 2 months post group completion
  30 item self-report scale that measures the phenomenology of the shame experience
World Health Organization Disability Assessment Schedule (WHODAS) to assess change between baseline, midpoint, group completion and 2 months post group. | Weeks 1, 4, 8 and 2 months post group completion
  12 item generic assessment instrument for health and disability

CONTACTS AND LOCATIONS:
Overall Officials: Rodelyn Wisco, MSW, Principal Investigator — Mount Sinai Hospital, Sinai Health System
Locations (1):
- Mount Sinai Hospital, Canada, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Gruber M, Hettema JM, Hwang I, Sampson N, Yonkers KA. Co-morbid major depression and generalized anxiety disorders in the National Comorbidity Survey follow-up. Psychol Med. 2008 Mar;38(3):365-74. doi: 10.1017/S0033291707002012. Epub 2007 Nov 30. PMID 18047766
- [Background] Patten SB, Gordon-Brown L, Meadows G. Simulation studies of age-specific lifetime major depression prevalence. BMC Psychiatry. 2010 Oct 20;10:85. doi: 10.1186/1471-244X-10-85. PMID 20961404
- [Background] Sundquist J, Lilja A, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Mindfulness group therapy in primary care patients with depression, anxiety and stress and adjustment disorders: randomised controlled trial. Br J Psychiatry. 2015 Feb;206(2):128-35. doi: 10.1192/bjp.bp.114.150243. Epub 2014 Nov 27. PMID 25431430
- [Background] Canadian Psychiatric Association. Clinical practice guidelines. Management of anxiety disorders. Can J Psychiatry. 2006 Jul;51(8 Suppl 2):9S-91S. No abstract available. PMID 16933543
- [Background] Parikh SV, Segal ZV, Grigoriadis S, Ravindran AV, Kennedy SH, Lam RW, Patten SB; Canadian Network for Mood and Anxiety Treatments (CANMAT). Canadian Network for Mood and Anxiety Treatments (CANMAT) clinical guidelines for the management of major depressive disorder in adults. II. Psychotherapy alone or in combination with antidepressant medication. J Affect Disord. 2009 Oct;117 Suppl 1:S15-25. doi: 10.1016/j.jad.2009.06.042. Epub 2009 Aug 13. PMID 19682749
- [Background] Teasdale JD, Cox SG. Dysphoria: self-devaluative and affective components in recovered depressed patients and never depressed controls. Psychol Med. 2001 Oct;31(7):1311-6. doi: 10.1017/s003329170100424x. PMID 11681557
- [Background] Gayner B, Esplen MJ, DeRoche P, Wong J, Bishop S, Kavanagh L, Butler K. A randomized controlled trial of mindfulness-based stress reduction to manage affective symptoms and improve quality of life in gay men living with HIV. J Behav Med. 2012 Jun;35(3):272-85. doi: 10.1007/s10865-011-9350-8. Epub 2011 May 20. PMID 21597980
- [Background] Germer CK, Neff KD. Self-compassion in clinical practice. J Clin Psychol. 2013 Aug;69(8):856-67. doi: 10.1002/jclp.22021. Epub 2013 Jun 17. PMID 23775511
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Spitzer RL, Williams JB, Kroenke K, Linzer M, deGruy FV 3rd, Hahn SR, Brody D, Johnson JG. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. JAMA. 1994 Dec 14;272(22):1749-56. PMID 7966923
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- See also: Centre for Addiction and Mental Health. Mental Illness and Addictions: Facts and Statistics — http://www.camh.ca/en/hospital/about_camh/newsroom/for_reporters/Pages/addictionmentalhealthstatistics.aspx
- See also: National Institute for Health and Care Excellence. Depression in adults: recognition and management. — http://www.nice.org.uk/guidance/cg90
- See also: WHO. WHO Disability Assessment Schedule 2.0 — http://www.who.int/classifications/icf/more_whodas/en/
- See also: Canadian Psychiatric Association and The College of Family Physicians of Canada — https://ww1.cpa-apc.org/Publications/Position_Papers/Shared.asp
- See also: Behavioral Medicine: A Primary Care Approach — https://books.google.ca/books?id=G0ITeV5CJYoC&pg=PA3&lpg=PA3&dq=80%25+primary+care+exclusive+mental+health&source=bl&ots=a1CDlNe1A3&sig=GWf-zOJ9V5fbmpFCpNAUl3qQy94&hl=en&sa=X&ved=0ahUKEwiYya3S-KjQAhVjqFQKHW0-DYgQ6AEILTAC#v=onepage&q=80%25%20primary%20care%20exclusive%20mental%20health&f=false